CLINICAL TRIAL: NCT00388388
Title: Double-blind, Randomized, Parallel Design Study Comparing Effectiveness of Losartan vs. Hydrochlorothiazide in Reversing or Preventing the Progression of the Remodeling of Resistance Arteries in Pre-hypertensive Pre-diabetic Subjects
Brief Title: Losartan Versus Hydrochlorothiazide in Reversing Remodeling of Small Arteries in Pre-Hypertensive Pre-Diabetic Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Few subjects recruited, sponsor withdrew support.
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Principal Investigator, Ernesto L. Schiffrin, Physician-in-Chief, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPC030
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Pre-hypertension; Pre-diabetes
Keywords: Remodeling; Resistance arteries; angiotensin receptor blocker; thiazide diuretic
MeSH Terms: conditions — Prehypertension; Glucose Intolerance | interventions — hydrochlorothiazide, losartan drug combination; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Losartan treatment
  Interventions: Drug: losartan, hydrochlorothiazide
- 2 (Active Comparator): Hydrochlorothiazide, 12.5-25 mg per day once a day for 6 months
  Interventions: Drug: losartan, hydrochlorothiazide

INTERVENTIONS:
Drug: losartan, hydrochlorothiazide — Losartan, 50-100 mg per day, once a day, for 6 months. Hydrochlorothiazide, 12.5-25 mg per day, once a day, for 6 months.
  Other Names: Cozaar, Apo-hydro

SUMMARY:
This randomized, double-blind, parallel group, two-centre pilot study will test the hypothesis that subjects who are otherwise healthy but fulfill the criteria for a diagnosis of pre-hypertension and pre-diabetes will have regression or reduced progression of hypertension-associated changes in their resistance arteries if their blood pressure is controlled for 6 months with losartan, whereas similar subjects whose blood pressure is equally well controlled using hydrochlorothiazide will have significantly less improvement of the changes in their resistance arteries.

DETAILED DESCRIPTION:
This randomized, double-blind, parallel group, two-centre pilot study will test the hypothesis that subjects who are otherwise healthy but fulfill the criteria for a diagnosis of pre-hypertension and pre-diabetes will have regression or reduced progression of hypertension-associated changes in their resistance arteries if their blood pressure is controlled for 6 months with losartan, whereas similar subjects whose blood pressure is equally well controlled using hydrochlorothiazide will have significantly less improvement of the changes in their resistance arteries.

The study will be conducted by Dr. Ernesto Schiffrin at the Cardiovascular Prevention Center, Sir Mortimer B. Davis Jewish General Hospital, McGill University, in Montreal, in association with a co-investigator at a second site, Dr. Rhian M. Touyz at the Ottawa General Hospital's Hypertension Clinic at the Riverside Campus and Kidney Research Center (University of Ottawa/Ottawa Health Research Institute). Over the past 15 years, Dr. Schiffrin has developed the gluteal subcutaneous biopsy methodology to be applied in the study. The technique has been practiced for many years (15 years) by Dr. Schiffrin, who more recently has collaborated with Dr. Touyz who used the technique together with Dr. Schiffrin before moving to Ottawa in 2005. In addition, stiffness of aorta (carotid-femoral pulse wave velocity) and endothelium-dependent hyperemic responses will be evaluated. Dr. Schiffrin and Dr. Touyz will be responsible for patient recruitment, data collection and analysis, and maintenance of study charts and patient records. Merck-Frosst Canada Ltd (MFCL) will be responsible for the study budget and the supply of medication.

The study subjects (men or women, 25 to 70 years of age) will be divided into two groups. Individuals with pre-hypertension (blood pressure = 120-139/85-90 mmHg) will be double-blindly allocated to either losartan or hydrochlorothiazide therapy respectively in groups 1 and 2. Study subjects will be assessed for their compatibility with inclusion and exclusion criteria, and subjects meeting the criteria will undergo baseline biopsies of gluteal subcutaneous resistance vessels. In addition, stiffness of aorta (carotid-femoral pulse wave velocity) and finger endothelium-dependent hyperemic responses will be evaluated. Subjects in each treatment group will receive antihypertensive therapy for 6 months, to control their blood pressure to 100-120/70-80 mmHg, and then have repeat gluteal biopsies, aortic stiffness and endothelial function measurements. The media/lumen ratio of resistance arteries 150-300 um in lumen diameter in the biopsied tissues will be determined. Previous work (1-3) has shown this parameter to be a useful marker of hypertensive vascular disease which may be modified by treatment with antihypertensive agents, particularly blockers of the renin-angiotensin system.

Subjects will give informed consent, and be medically assessed to determine whether they satisfy the inclusion and exclusion criteria. Eligible subjects will have a sitting systolic blood pressure (SiSBP) 120-139 mmHg, and be otherwise in good health. Eligible subjects will have a gluteal biopsy, and then be randomized to treatment group 1 or group 2 for 6 months.

For study purposes, SiSBP will be defined as the average of three consecutive valid readings, taken at one-minute intervals after five minutes of repose.

Thirty subjects who satisfy the study criteria will be randomized to receive once daily therapy with either losartan 50 mg or hydrochlorothiazide 12.5 mg. Subjects will take study medication once daily between 06:30 and 11:00, and be followed up in morning clinic visits, scheduled between 06:30 and 11:00. Subjects will be instructed not to take their medication on the morning of clinic visits until after the clinic evaluations have been completed. During the 6 months of treatment, subjects will have their "trough" blood pressure, heart rate (HR) and body weight measured at every clinic visit. At visits where laboratory safety tests will be done, subjects will be asked to come fasting.

All subjects will be force-titrated to losartan 100mg daily or hydrochlorothiazide 25 mg daily. However, if they develop dizziness and/or SiBPs below 100/70 mmHg, the dose may be down-titrated back to 50 mg losartan or 12.5 mg hydrochlorothiazide.

If any subjects develops SiBPs > 139/90 mmHg, open label amlodipine will be give to maintain SiBP < 139/90 mmHg, attempting however to reach the goal of SiSBP < 120 mmHg. Amlodipine will be started at a dose of 2.5mg daily and up-titrated every 4 weeks to 5 mg daily and then to 10 mg daily. As long as SiBP < 139/90 mmHg, subjects will not be discontinued from the study. Subjects whose hypertension is not adequately controlled (SiBP > 139/90 mmHg) with addition of amlodipine up-titrated to 10 mg daily, however, will be discontinued from the study.

Laboratory safety tests will be done at Weeks 4, 12, 24 of double-blind therapy (Visits 6, 8 and 9). An ECG will be repeated at the end of the study (Week 24).

The study will start at the end of 2006, last approximately 1 year. Recruitment should be completed within 6-9 months. Duration of other periods has been specified briefly above within the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Prehypertensive prediabetic subjects (25-70 years old) defined as otherwise normal subjects with a mean SiSBP of 120-139 mmHg and fasting blood glucose of 6.1-6.9 mmol/L or impaired glucose tolerance on oral glucose tolerance test (OGTT) at screening and after two weeks of placebo therapy (Week -2)

Exclusion Criteria:

* Hypertension or clinically significant renal disease
* Cerebrovascular accident within the past year, or current transient ischemic attacks
* Myocardial infarction within the past year; percutaneous coronary angioplasty or coronary artery bypass surgery within last 6 months
* Clinically significant AV conduction disturbances and/or arrhythmias (e.g. second- or third-degree AV block; sick-sinus syndrome or clinically significant bradycardia- resting heart rate < 45 beats/minute), tachyarrhythmias; clinically significant arrhythmias, presence of accessory bypass tract (e.g. Wolff-Parkinson-White syndrome)
* Angina pectoris
* Current or prior history of heart failure or known left ventricular ejection fraction <40%
* History of unexplained syncope or known syncopal disorder (e.g., Stokes-Adams Syndrome)
* Known history of hemodynamically significant obstructive valvular disease or hypertrophic cardiomyopathy
* Use of agents that may cause alteration of blood pressure is prohibited. This includes nitrates, or alpha or beta-blockers. Calcium channel blockers are allowed as second line therapy if hypertension develops during the study Major psychotropic agents and antidepressants are not permitted
* Cimetidine is not permitted (famotidine and ranitidine and proton pump inhibitors are allowed).
* NSAIDs are permitted if taken on a stable regimen. Aspirin in small doses (< 1 g/day) as cardioprotective agent and acetaminophen are permitted
* Oral or inhaled steroids, ACTH, immunosuppressants or lithium are not allowed
* Serum creatinine concentration >200 μmol/L (adjusted for age and weight)
* Urine dipstick or microscopic findings suggestive of significant renal or other disease.
* Hematuria should be evaluated, the etiology established/documented, and treatment rendered as appropriate prior to entry
* Off-treatment serum potassium concentration >5.5 mmol/L or <3.5 mmol/L
* AST (SGOT) or ALT (SGPT) >2 x normal upper limit
* Clinically significant laboratory values outside of the established normal range including but not limited to the following parameters: hemoglobin, platelet count or white blood cell count
* Known hypersensitivity or contraindication to losartan or thiazide diuretics
* History of clinically important malabsorption or gastrointestinal resection
* Current urinary tract infection
* Smoking 10 cigarettes or more.
* Pregnancy or lactating females. Females of childbearing age who are not surgically sterilized and are using effective contraception may enter only if an exclusionary pregnancy test is done within 72 hours of the first double-blind dose of test agent. Pregnancy tests will then be done monthly throughout the study.
* Vasculitis or vasculopathy: collagen-vascular diseases, chronic hepatitis B antigenemia, circulating immune complexes, complement disorders, amyloidosis, scleroderma, etc. Neoplasms, Acquired Immunodeficiency Syndrome (AIDS), or HIV positive
* Bleeding or platelet disorder
* Known absence of one kidney
* Subjects abusing or who within past two years abused alcohol or other drug substances
* Mentally or legally incapacitated subjects
* Subjects who have participated in another investigational drug trial, including those using marketed drugs (i.e. patient has signed a consent form), within the 28 days prior to start of placebo therapy
* Subjects who, in the opinion of the investigator, will not cooperate fully, keep appointments or are unreliable
* Inability or unwillingness to sign the Patient Consent Form
* Phase V of Korotkoff sounds cannot be detected

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Effect of 6 months of losartan or hydrochlorothiazide on media/lumen ratio of gluteal subcutaneous resistance arteries in otherwise normal subjects who fulfill criteria for pre-hypertension and pre-diabetes | 6 months

SECONDARY OUTCOMES:
Safety and tolerability of 6 month therapy with losartan or hydrochlorothiazide, and effect on media thickness, lumen diameter and vascular function of gluteal subcutaneous resistance arteries, and serum and tissue inflammatory markers in same subjects | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto L. Schiffrin, MD, PhD, Principal Investigator — Physician-Chief, SMBD - Jewish General Hospital & Professor of Medicine, McGill University
Locations (1):
- Cardiovascular Prevention Centre, Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Schiffrin EL, Park JB, Intengan HD, Touyz RM. Correction of arterial structure and endothelial dysfunction in human essential hypertension by the angiotensin receptor antagonist losartan. Circulation. 2000 Apr 11;101(14):1653-9. doi: 10.1161/01.cir.101.14.1653. PMID 10758046
- [Background] Park JB, Intengan HD, Schiffrin EL. Reduction of resistance artery stiffness by treatment with the AT(1)-receptor antagonist losartan in essential hypertension. J Renin Angiotensin Aldosterone Syst. 2000 Mar;1(1):40-5. doi: 10.3317/jraas.2000.009. PMID 11967798
- [Background] Schiffrin EL, Park JB, Pu Q. Effect of crossing over hypertensive patients from a beta-blocker to an angiotensin receptor antagonist on resistance artery structure and on endothelial function. J Hypertens. 2002 Jan;20(1):71-8. doi: 10.1097/00004872-200201000-00011. PMID 11791028
- [Background] Savoia C, Touyz RM, Endemann DH, Pu Q, Ko EA, De Ciuceis C, Schiffrin EL. Angiotensin receptor blocker added to previous antihypertensive agents on arteries of diabetic hypertensive patients. Hypertension. 2006 Aug;48(2):271-7. doi: 10.1161/01.HYP.0000230234.84356.36. Epub 2006 Jun 19. PMID 16785331
- See also: Sir Mortimer B. Davis - Jewish General Hospital and Lady Davis Institute for Medical Research — http://www.jgh.ca